# The effect of intensive hipotherapy on the psychomotoric development of children with spinal muscular atrophy (HIPOSMA)

### 1. Introduction

Spinal muscular atrophy is rare neuromuscular disease, it is caused by gene mutation SMN1. This gene encodes SMN protein. This protein is most important to survive alfa-motoric neurons in spinal cord. When this protein doesn't work, no signals go from brain to skeletal muscles and fazic muscles of body. In the end weakening breathing muscles and internal organs muscles. The first treatment is pharmacological treatment. There is a lot of research about medicament treatment, the famous treatment in Czech Republic is medicine Spinraze and from year 2020 medicine Zongelsma. This, however, more often puts more difficulty on complex rehabilitation. An empirical observation has found out that complex rehabilition has positive effect on progress of disease and on self-sufficiency of people and children with SMA. Physiotherapy is one of the recommended rehabilitation types.

The use of rehabilitation procedures is common in clinical practice. In a 2016 study, 105 adults with SMA were asked how many of them used physiotherapy. A total of 86% of respondents received these services, yet the authors of the article conclude that further research is needed to understand the impact of physiotherapy in SMA.

Nevertheless, there is a lot of discussion if physiotherapy is really good for people and children with SMA. Some research shows us, that physiotherapy doesn't worsen this disease. Lewelt et al. in their research they showed that strength training 3 times a week does not show side effects in children under 10 years of age, in some cases trends in improving muscle strength and motor functions have been observed.

Because in physiotherapy we work primarily with muscles, and a lot of activity can cause fatigue of skeletal muscles and worsen their function. But from clinical work we know that the effect of physiotherapy is extensive. There is a research on mice which shows the effect of physiotherapy on the strength activities and the aerobic activities.

Research to better elucidate the intensity of physiotherapy has not yet been published. Motes et al. monitored a total of 16 patients with SMA aged 10 - 55 years, who regularly underwent home autotherapy for 16 months - cycling and strengthening. The authors did not find any side effects of exercise on strength, function or fatigue during the study. However, the

oxidation capacity has been reduced and according to the authors, further research is needed in this area.

In the United States, the "Standard of Care" (SMA-SOC) has been developed for SMA, which regulates the rehabilitation care of children and adults with SMA according to the degree of mobility. In the framework of the said directive, the stretching of contractures, swimming, water therapy, light strength exercises and a verticalization stand are recommended within the framework of physiotherapy, and horse riding is also mentioned - but without more detailed information. Vibration techniques and positioning are recommended to improve breathing. Recommended exercises for seated persons also include concentric and eccentric exercises and aerobic and general fitness exercises with and without resistance. According to the directive, the duration of therapy should be adapted to the individual patient. For walkers, the exercise program may include some forms of balance exercises, dynamic and static.

In a study from 2021, physiotherapists were asked about their knowledge of SMA-SOC and its use in practice. Most of them stated that after individuals with SMA started disease-modifying pharmacotherapy, they would recommend increasing the frequency and duration of therapeutic interventions. The authors agree that in practice there are differences in the care of people with SMA, especially in the frequency and duration of specific interventions. At the same time, they state that these findings can identify future research needs and thus extend SMA-SOC to rehabilitation management best practices

Our goal is to compare two physiotherapeutic approaches - the recommended form of classical physiotherapy and the method on a neurophysiological basis - hippotherapy. Due to the nature of the disease, we expect a greater effect in the method of Hippotherapy in DMO, where several muscle chains work simultaneously and thus succeeds in activating weakened muscles within the chain, which eliminates possible fatigue and worsening of the condition. However, we also expect a positive effect in the recommended form of classical physiotherapy. Here, however, due to the lower intensity of the sensory environment and the possible complexity of movement, we assume less effectiveness than hippotherapy.

The secondary intention of the research will be the appropriate intensity of therapy so that unwanted muscle fatigue does not occur. We will therefore investigate the neurophysiological mechanisms of rehabilitation that we will monitor using long non-coding RNAs (lncRNAs)

involved in important cellular regulation, including regulation of genomic imprinting, epigenetic chromatin modification, transcriptional interference, and nuclear export. The lncRNA, SMN-antisense 1 (SMN-AS1), has been shown to repress the expression of the duplicate SMN2 gene by binding Polycomb repressive complex 2 (PRC2) to its locus. Increasing the transcriptional activity of an almost identical SMN2 gene can functionally compensate for the loss of SMN1, increase the amount of SMN protein and thus improve the prognosis of the disease. Chemically modified oligonucleotides have been proposed that disrupt the interaction between SMN-AS1 and PRC2, which inhibits the action of PRC2 and thus leads to increased SMN2 expression. (Woo C J et al.) Investigation of lncRNAs involved in the processes of gene regulation of these genes may help to understand the neurophysiological effects of rehabilitation of children with SMA.

# 2. Participants and method

### a. Clinical trial design

In randomized controlled study will compare 2 groups of children, in ages 1 - 8 years old. First group will have physiotherapy on the neurophysical basis. It will last 6 days with intensity once a day cca 30 minutes. Second group will have hippotherapy, it will last 6 days too. Hippotherapy will be twice a day, cca 15 minutes.

Both forms of physiotherapy will focus on psychomotoric development of children and on improvement stability and gross motoric function. Both groups will have one more therapy, especially therapeutic grooming. Goals of this activity is improvement of psychosocial development of children. All children will be evaluated before and after rehabilitation intervention.

### b. Eligibility criteria

Inclusion criteria: clinic diagnosis SMA (I, II, and III types), children's age 1-8 years, no changing medicine 6 months at least, without another grave diseases

Exclusion criteria: hip subluxation, allergies to horses and the environment of horse stables, insurmountable fear of the horse

# c. A detailed description of two groups

Both groups will have 6 days long therapeutic programm (in same length and intesity) -1 of day 15 minutes intensive therapy plus 1 a day therapeutic grooming 20 minutes long, with same therapeutic goal. For practical reasons, classical physiotherapy will be performed in a common block - i.e once a day for 30 minutes.

Both forms physiotherapy will develope psychomotoric development of children, motorskills, mobility and independent, stability and symmetry. Therapeutic grooming will develop psychosocial development of children.

Therapeutic grooming: In order to influence the psychomotor development in a comprehensive way, the psychosocial activity of therapeutic grooming will also be included in the study. Its goal is to support children's communication, their interaction with the environment, the ability to establish contact with the horse and the overall emotional support of children with SMA. The purpose of this activity is to clean the horse, its possible guide, stroking and contact with the horse, work from the ground.

# **Group 1: Individual physiotherapy (SMA-SOC)**

Therapeutic procedures according to the recommended standard (SMA-SOC) will be used in the therapy. Elements of breathing gymnastics, vibration techniques, stretching, eccentric and concentric exercise procedures will be combined. Individual physiotherapy will be conducted on the basis of set goals from the kinesiological examination, it will be adapted to the individuality of the child - his cooperation, fatigue and sleep time.

### Group 2: Hippotherapy by the children with cereberal palsy (HT by CP)

HT by CP is an accredited form of hippotherapy, whose methodology is based on the clinical picture of cereberal palsy, but its procedures are applicable to a wider group of children with disabilities. Therefore, we anticipate its effect for children with SMA. Based on a special type of examination, this method precisely determines the "type / breed" of the horse according to the biomechanics of the movement of its back in the step, the position of the child and the neurophysiological function of the back - differentiation or sensorimotor skills. Furthermore, according to the course of therapy, the physiotherapist determines the pace of the horse's step, its length, selects special manual contacts according to the current situation and adjusts the duration of therapy to the client's fatigue. Therapy will be performed by therapists with professional competence to perform hippotherapy by children with CP.

# d. Pre- and post-intervention assessments

In study will give the participants this basic datas – age and gender, information about disease: time, who the diagnosis was determinated, beginning of medicament treatment, until rehabilitation, current pharmacological treatment, if the child has some pains, use of compensatory aids, maximum possible independence of the child, presence and current state of a scoliosis, current motoric and physical activity of child

Clinic and instrument observation will be 1 -1,5 hours long. All these will be adapted to children's sleeping patterns and fatiques. Both observation will be very difficult. For this reason there will be a game prepared, with some treasure at the end.. In the end became treasure.

### e. Outcomes and measures

### **Primary outcomes:**

### 1. The ability of the thorax to change shape

The examination will take place lying on your back. 3 position markers will be placed on each side of the thorax, in the area of the distal end of the sternum axes, at the level of the 3rd rib and at the lowest arch of the 10th rib. Their position during exhalation and inspiration will be measured, and the change in thorax circumference will be evaluated. The aim of this test is to objectify the change in respiratory stereotype. After therapy, we expect a greater ability of the thorax to change direction.

# 2. Sitting symmetry

Observations will be made by sitting on a therapy cylinder. There will be special markers on the body (on clothes) of children: lower angles of the scapulae axes, ridge of the iliac axes, sacroiliac joint (SI) on both sides and in the area of the L4 vertebra and navel. We will measure the symmetry of these marks in each other's position and the movement in which the

child will walk back and forth with his hands. Markers will be analyzed using Qualisys Motion Capture Systems 2020.3. Acceleration and change of position will be evaluated in the second time.

# 3. Work with the center of gravity

Observation will be performed by sitting on therapeutic cylinder. 3 position markers will be used on each side of the body, at the root of the palm, in the area of the SI joint and at the level of the temporomandibular joint. The change of markers will be measured from the starting position until the child is stretched to the side (torso tilt with lug) and forward (torso flexion with forearm). The monitoring child will be motivated to reach for a toy. The goal is to evaluate the stability of children. We assume, that after therapy we can see better work with the center of gravity.

### 4. Muscle fatigue

We will measure muscle fatigue after physical activity using surgace EMG. The child will lie on its back, therapist will provide a toy in the area of his opposite knee. The child will stretch for this toy. This act will take 30 s. We will evaluate activity m. obliquus externus abdominis at the beginning and end of this specific activity. Goal is to evaluate muscle fatigue. We assume that after the intensive therapeutic program the muscle fatigue will be lower.

# 5. Hammersmith function scale for children with spinal muscular atrophy

The examination will follow a standardized procedure.

# 6. Deep neck flexor endurance test

We assume that after an intensive rehabilitation we will see better qualitative activity deep neck flexor.

### 7. Neck extensor endurance test

We assume that after an intensive rehabilitation we will see better qualitative activity neck extensor.

### 8. Spirometric measure

The spirometer will be used to determine the FEV1 value, i.e the volume of air exhaled after the maximum inspiration with the greatest effort within 1 second. The change in value at the beginning and end of the rehabilitation stay will be evaluated.

# The secundary outcomes:

# 9. Quality of life

Parents of child with SMA will fill special questionnaire at the beginning and two weeks after end of the rehabilitation. The ICF score set, more precisely the ICF-based Documentation Form, the category Children with cereberal palsy Brief (below 6 years old), supplemented by some items from the rehabilitation set, will be used to evaluate the quality of life.

# 10. Monitoring of molecular biological indicators of rehabilitation

All blood will be taken on an empty stomach for RNA analysis. The A RiboPure TM -Blood Kit (cat # AM1928, ThermoFisher Scientific) will be used to isolate high quality RNA directly from all the blood. This kit contains RNAlater® Solution (cat. # AM7020, ThermoFisher Scientific), which protects RNA and is designed to allow later processing of samples (not immediately after sampling), which is more processable. RNAlater® Solution also blocks a given cell gene expression profile. Samples treated in this way can be safely stored at room temperature for longer periods of time (up to three days or more). Blood samples stored in RNAlater® Solution achieve RNA quality comparable to the quality of samples processed immediately according to commercial websites. The expected average total RNA yields will be about 2-4 g / 0.5 ml of all blood. Total RNA will be transcribed into cDNA by reverse transcriptase. To avoid error, the expression of human lncRNA and internal endogenous gene (e.g., GAPDH) will be quantified using RNA obtained from blinded samples (i.e., concealment of sample origin allocation).

Blood collection will always take place in the morning before and after the complete end of the rehabilitation course, directly at the place of accommodation of families with children with SMA.

# 3. Hypotheses

This clinical trial will test the following scientific hypotheses:

1. We assume *that even* if both of the therapies are so intesive, there is no unwanted muscle fatigue.

Hippotherapy is 15 minutes long, twice a day, classic physiotherapy 30 minutes ones a day. Of course, all therapies will be adapted to children's fatique. The goal of therapies is to stimulate physiological muscle interactions and to eliminate unilateral loading of individual muscles. In the second case inappropriate overload is too dangerous.

2. We assume that these tests: work with the center of gravity, sitting symmetry and the ability of the thorax to change shape there will be a significant improvement in the second group (*hippotherapy*).

During hippotherapy child must respond to slight deviations of the horse's back, these deviations stimulate work with the center of gravity and in the second time breathing stereotype. The walk of horses are rythmic and periodic. The answer the child's motor skills is symmetric differentiation. We hope, that symmetric differentiation has a major effect on the symmetry of the sitting.

3. We assume, that *hippotherapy* (group 2) will have better effect than *classic* physiotherapy (group 1) by the tests: work with the center of gravity and sitting symmetry.

The horseback movement stimulates symmetric differentiation and activation of the deep muscles of the spine. Both in hight intesity.

4. We don't assume there will be significant improvement by the test HFS.

The test HFS has low sensitivity and records quantitative change rather than qualitative changes.

5. We assume there will be significant improvement by the parameter FEV1 (spirometric measurement). This improvement will be by both therapeutic concept.

It's very important to make therapies of diaphragm area. In hippotherapy, what helps us is the horseback movement in transverse plane, in physiotherapy we work with breathing exercise. These will cause a targeted effect on the diaphragm area.

6. We assume there will be significant improvement by the group 1 (classic physiotherapy) by these tests: Deep neck flexor a neck extensor endurance test.

In classic physitoherapy we can local stimulate deep neck flexor and neck extensor. Equally, we hope for a significant improvement.

# **Informed Consent Form (in Czech)**

# Informace pro pacienta

Vážený pane/vážená paní,

Vyzýváme Vás a Vaše dítě k účasti na vědecké studii, jejímž cílem je ověřit efektivitu intenzivní fyzioterapie u dětí se spinální muskulární atrofií. Studie bude probíhat v rámci 6ti denního rehabilitačního programu, jehož náplní bude hipoterapie či individuální fyzioterapie.

Přečtěte si prosím informace o studii a rozhodněte se, zda máte zájem se se svým dítětem do výzkumu zapojit.

Věřím, že Vás tato možnost zaujme.

Mgr. Kateřina Maříková, CH Mirákl, o.p.s., Bohuslavice, hlavní řešitel studie

# Informace pro pacienta

# a) Název studie:

Vliv intenzivní hipoterapie na psychomotorický vývoj dětí se spinální svalovou atrofií

b) V rámci studie vám bude rehabilitační program nabídnut zcela zdarma. V současné době je žádáno o finanční podporu nadaci TKH pro příspěvek na ubytování rodin účastnících se studie.

c) Hlavním řešitelem studie je Mgr. Kateřina Maříková:

Centrum hiporehabilitace Mirákl, o.p.s., Bohuslavice 10, Telč 58856, IČ 2290567

Email: katerina.marikova@chmirakl.cz

Telefon: 607616104

d) Plánovaný počet účastníků studie

Plánujeme, že během jednoho roku se uskuteční dva rehabilitační pobyty s celkovým počtem 16ti dětí.

e) Účel studie

Cílem studie je ověření významu intenzivní fyzioterapie pro děti s SMA a srovnání dvou terapeutických konceptů, postavených na aktivaci fyziologických svalových souher v krátkém časovém úseku, ale v intenzivní formě tak, aby výsledkem bylo celkové zlepšení samostatnosti dítěte a kvalitativní zlepšení psychomotorického vývoje. Terapeutickými koncepty budou hipoterapie a individuální fyzioterapie.

f) Popis výzkumných procedur

# Organizace studie

V randomizované kontrolované studii budou porovnávány dva fyzioterapeutické koncepty u dětí s SMA ve věku 2-8 let, schopné samostatného sedu. Obě skupiny podstoupí šestidenní terapeutický program stejné délky a intenzity (2x denně 15 min. individuální terapie + 1x denně 20 min. terapeutické čištění koní) se stejným terapeutickým cílem.

Jedna skupina podstoupí fyzioterapii dle doporučovaných směrnic SMA-SOC, druhá hipoterapii. Primární výstupy budou vyšetřeny před začátkem a na konci terapeutického programu (Test schopnosti hrudníku měnit tvar, symetrie sedu, schopnosti práce s těžištěm, unavitelnosti svalů, vzniku kontraktur; Hammersmithova funkční škála pro děti se spinální muskulární atrofií, vyšetření krve, Deep neck flexor and Neck extensor endurance test). Sekundární výstupy budou vyšetřeny před a 5 týdnů po ukončení programu (dotazník kvality života).

### Účastníci studie

Kritéria pro zahrnutí do studie:

- klinická diagnóza SMA (I, II i III typu)
- věk 2-8 let
- schopnost samostatného sedu
- s neměnnou medikací alespoň 6 měsíců
- bez dalších vážných přidružených onemocnění

# Vylučující kritéria:

- subluxace kyčelních kloubů
- alergie na koně a prostředí koňských stájí nepřekonatelný strach z koně

# Základní údaje

Ve studii budou účastníci uvádět základní sociodemografické (věk, pohlaví) a anamnestické údaje: doba určení diagnózy onemocnění (potvrzená délka onemocnění), začátek a typ medikace (délka medikace) a současná farmakologická léčba, přítomnost bolesti, dosavadní rehabilitace, užívání kompenzačních pomůcek, maximální možná samostatnost dítěte, přítomnost a současný stav skoliózy, současná aktivita dítěte motorická i psychická.

# Fyzioterapeutické vyšetření

Přístrojové i klinické vyšetření bude trvat přibližně 1-1,5 hodiny. Doba vyšetření bude přizpůsobena spánku dítěte a jeho spolupráci. Z důvodu časové náročnosti vyšetření bude pro děti vymyšlena hra, ve které budou plnit jednotlivé úkoly v podobě vyšetření s cílem získat "poklad".

### Primární výstupy

V biomedicínské laboratoři na Vysoké škole polytechnické v Jihlavě budou měřeny následující testy:

# 1. Schopnost hrudníku měnit tvar

Vyšetření proběhne v sedu na válci. Na hrudníku budou umístěny polohové markery, a to v oblasti processus styloideus, na úrovni 4. žebra bilaterálně, distálním konci klíční kosti bilaterálně, na vrcholu oblouku 10. žebra, vztahovat se budou k markeru v oblasti C7 a thorakolumbálního přechodu. Markery budou umístěny na přiléhavém oblečení dětí. Měřeno bude jejich postavení při výdechu a nádechu, hodnocena pak změna obvodu hrudníku. Cílem tohoto testu je zaznamenat změnu dechového stereotypu. Po terapii předpokládáme větší schopnost hrudníku měnit směr.

### 2. Symetrie sedu

Vyšetření proběhne v sedu na válci. Na přiléhavém oblečení dětí bude umístěno několik polohových markerů: dolní úhly os scapulae, hřeben os iliaca, sacroiliakální skloubení (bilaterálně), a v oblasti obratle L4 a umbilicus. Děti budou pohybovat rukami po válci dopředu a zpět. Měřena bude vzdálenost markerů od páteře, hodnocena pak jejich symetrie ve vzájemném postavení. Markery budou zaznamenány pomocí Qualisys Motion Capture Systems 2020.3. Následně bude vyhodnoceno zrychlení a změna polohy.

### 3. Schopnost práce s těžištěm

Vyšetření proběhne v sedu na válci. Na každé straně těla budou použity 3 polohové markery, na kořenu dlaně, v oblasti SI skloubení a na úrovni temporomandibulárního kloubu. Měřena bude změna markerů z výchozí pozice do natažení dítěte do strany (úklon trupu s upažením) a dopředu (flexe trupu s předpažením). Dítě bude motivováno, aby se natáhlo po hračce. Cílem je posoudit stabilitu dětí, kdy po terapii předpokládáme větší schopnost vychýlení z těžiště.

### 4. Unavitelnost svalů

Pomocí povrchového EMG bude měřena unavitelnost svalů po fyzické aktivitě. Dítě bude ležet na zádech, terapeut mu bude v oblasti jeho protilehlého kolena nabízet hračku, pro kterou se bude dítě natahovat. To vše po dobu 30 s. Měřena bude aktivita m. obliquus externus abdominis na začátku a na konci této specifické aktivity. Cílem je zhodnotit unavitelnost svalů. Očekáváme, že po ukončení intenzivní rehabilitace bude unavitelnost svalu nižší.

Na pracovišti CH Mirákl budou vyšetřeny tyto validované testy:

**1.** Hammersmithova funkční škála pro děti se spinální muskulární atrofií Vyšetření proběhne dle standardizovaného postupu.

# 2. Deep neck flexor endurance test

Očekáváme kvantitativní zlepšení v tomto testu ve smyslu kvalitnějšího zapojení hlubokých flexorů krku po intenzivní rehabilitaci.

### 3. Neck extensor endurance test

Očekáváme kvantitativní zlepšení v tomto testu ve smyslu kvalitnějšího zapojení extenzorů krku a páteře po intenzivní rehabilitaci.

# 3. Spirometrické měření

Pomocí spirometru bude zjišťována hodnota FEV1, tedy objem vzduchu vydechnutý po maximálním nádechu s největším úsilím během 1 sekundy. Hodnocena bude změna hodnoty na začátku a konci rehabilitačního pobytu.

# Sekundární výstupy

### Vvšetření kvality života

Rodiče či zákonní zástupci budou požádáni o vyplnění dotazníku na začátku studie a 4 týdny po ukončení rehabilitačního programu. Pro hodnocení kvality života bude využit ICF score set, přesněji ICF-based Documentation Form, kategorie Children with cereberal palsy Brief (below 6 years age old). (20)

### Monitorování molekulárně biologických ukazatelů rehabilitace

Pro analýzu RNA bude odebrána plná krev na lačno. Pro izolaci vysoce kvalitní RNA přímo z plné krve bude použit A RiboPure<sup>TM</sup>-Blood Kit (cat# AM1928, ThermoFisher Scientific). Tento kit obsahuje RNA*later*® Solution (cat.# AM7020, ThermoFisher Scientific), který chrání RNA a je navržen tak, aby umožnil pozdější zpracování vzorků (nikoliv hned po odběru vzorků), což je procesně lépe realizovatelné. RNA*later*® Solution také zablokuje daný profil genové exprese buněk. Takto ošetřené vzorky mohou být bezpečně skladovány při pokojové teplotě po delší časová období (až tři dny i více). Krevní vzorky skladované v

RNA*later*® Solution dosahují kvality RNA srovnatelné s kvalitou vzorků, zpracovaných okamžitě dle komerčních webových stránek. Očekávané průměrné výtěžky celkové RNA budou asi 2–4 μg/0.5 ml plné krve. Celková RNA bude reverzní transkriptázou přepsána do cDNA. Aby se předešlo chybě, bude exprese lidské lncRNA a interního endogenního genu (např. *GAPDH*) kvantifikována pomocí RNA získané ze zaslepených vzorků (to znamená utajení alokace původu vzorku).

Odběr krve proběhne vždy ráno před začátkem a po úplném skončení rehabilitační kůry, přímo v místě ubytování rodin s dětmi s SMA.

# **Terapie**

Obě skupiny podstoupí šestidenní terapeutický program stejné délky a intenzity (2x denně 15 min. individuální terapie + 1x denně 20 min. terapeutické čištění koní) se stejným terapeutickým cílem. Z praktických důvodů bude klasická fyzioterapie prováděna ve společném bloku – tedy 1x denně 30 minut.

Obě formy individuální fyzioterapie budou zaměřeny na podporu psychomotorického vývoje dětí, na rozvoj jejich hrubé motoriky a tím mobility a samostatnosti, na podporu stability a symetrie. Doplněná skupinová aktivita terapeutické čištění koní bude cílená na psychosociální rozvoj dětí.

# 1. skupina – individuální fyzioterapie (SMA-SOC)

V terapii budou využívané terapeutické postupy dle doporučovaného standardu (SMA-SOC) (4). Kombinovány budou prvky dechové gymnastiky, vibrační techniky, strečink, excentrické i koncentrické cvičební postupy. Individuální fyzioterapie bude vedena na základě stanovených cílů z kineziologického vyšetření, bude přizpůsobena individualitě dítěte – jeho spolupráci, únavě a době spánku. Terapii budou vykonávat fyzioterapeuti dle zákona 96/2004 Sb. Specializace ve zdravotnictví, Fyzioterapie pro držitele osvědčení fyzioterapeut a ergoterapeut.

# 2. skupina – Hipoterapie u DMO

Hipoterapie u DMO je akreditovaná forma hipoterapie, jejíž metodika je postavena na klinickém obraze DMO, ale její postupy jsou využitelné pro širší skupinu dětí se zdravotním znevýhodněním. Proto předpokládáme její efekt právě pro děti s SMA.

Tato metoda přesně stanovuje na základě speciálního typu vyšetření "typ/plemeno" koně dle biomechaniky pohybu jeho hřbetu v kroku, polohu dítěte a neurofyziologickou funkci hřbetu – diferenciaci či senzomotoriku. Dále dle průběhu terapie fyzioterapeut stanovuje tempo kroku koně, jeho délku, vybírá dle aktuální situace speciální manuální kontakty a přizpůsobuje délku terapie únavě klienta.

Terapii budou vykonávat terapeuti s odbornou způsobilostí pro výkon Hipoterapie u DMO.

# Terapeutické čištění koní

Pro možnost ovlivnění psychomotorického vývoje komplexně bude do studie zařazena i psychosociální aktivita terapeutické čištění koní. Jejím cílem je podpora komunikace dětí, jejich interakce s okolím, schopnost navázat kontakt s koněm a celková emoční podpora dětí s SMA. Náplní této aktivity je čištění koně, jeho možné vodění, hlazení a kontaktování se s koněm, práce ze země.

# g) Rizika účasti ve studii

Tato studie neskýtá žádná rizika. Vyšetření budou provádět kompetentní vyšetřující a terapii kvalifikovaní fyzioterapeuti.

### h) Přínos účasti ve studii

Účast ve studii Vám poskytne nadstandardní terapeutický přístup ve všech kohortách. Po ukončení studie obdržíte hodnocení výsledků vašeho dítěte, na vyžádání dostanete také závěrečnou zprávu o výsledcích této studie. Účastí na studii přispějete ke zvýšení efektivity rehabilitační péče o děti se spinální muskulární atrofií.

# i) Důvěrnost získaných informací

Vaše osobní data a data vašeho dítěte nebudou předávána žádné třetí osobě. Všechny vaše osobní údaje, i vašeho dítěte, budou uchovávány v papírové i elektronické podobě a hlavní zkoušející s jeho spolupracovníky budou se získanými daty nakládat v souladu s platnými zákony České republiky o ochraně osobních údajů. Vaše údaje budou v naší databázi anonymizovány, tj. budou odstraněny veškeré informace, které mohou být osobně identifikovatelné. Údaje budou i nadále uschovány pod zvláštním kódem a klíč pro dešifrování bude znám pouze hlavnímu zkoušejícímu. Lékařskou dokumentaci vašeho dítěte bude mít k dispozici pouze hlavní zkoušející a jeho spolupracovníci v týmu. K dokumentaci vašeho dítěte mohou mít přístup také zástupci schvalující etické komise.

### i) Kompenzace účasti

Účast na studii je plně dobrovolná a není nikterak honorována.

Účast na studii nemá žádná známá rizika, přesto v případně eventuálního poškození pokusné osoby související s její účastí na projektu, bude osoba kompenzována pojištěním organizace.

k) Adresy instituce a osob nezávislých na výzkumném projektu, které Vám mohou poskytnout informace o Vašich právech i o samotném výzkumném projektu:

Etická komise při Institutu klinické a experimentální medicíny a Thomayerově nemocnici

Vídeňská 800, 140 59 Praha 4

Kromě toho máte právo podat stížnost na způsob nakládání s vašimi údaji a můžete je zaslat příslušnému orgánu odpovědnému na provádění zákona o ochraně osobních údajů – Úřad pro ochranu osobních údajů se sídlem v Praze.

1) Podepsání informovaného souhlasu

Účast vašeho dítěte na studii je plně dobrovolná a můžete kdykoliv od tohoto rozhodnutí ustoupit.

Tento formulář je podepsán ve dvou originálech, z nichž jeden je pro Vás a druhý je uložen ve studijním centru.

Přečetl/a jsem si informace obsažené v tomto informovaném souhlasu. Měl/a jsem dostatek času přemýšlet o účelu, postupech, možných rizicích a výhodách účasti ve studii. Obdržel/a jsem uspokojivé odpovědi na všechny své otázky a věřím, že chápu všechny informace uvedené v tomto informovaném souhlasu.

Souhlasím s tím, že se budu řídit pokyny lékaře a budu jej okamžitě informovat o jakýchkoli nežádoucích účincích. Podpisem tohoto informovaného souhlasu se nevzdávám žádného ze svých zákonných práv.

Souhlasím se shromažďováním, používáním a zveřejňováním lékařských informací mého dítěte způsobem popsaným v tomto informovaném souhlasu.

# m) Ujištění

Ujišťujeme Vás, že budete včas informován/a o nově zjištěných okolnostech, které by mohly mít vliv na Vaše rozhodnutí v pokračování ve studii.

Účastník:

Jméno a příjmení tiskacími písmeny

Podpis:

# Informovaný souhlas

Název a popis studie: Vliv intenzivní hipoterapie na psychomotorický vývoj dětí se spinální svalovou atrofií

Jméno pacienta:

Datum narození:

Jméno zákonného zástupce:

Pacient byl do studie zařazen pod číslem:

Odpovědný lékař:

- 1. Já, níže podepsaný (á) souhlasím s účastí mého dítěte ve studii. Je mi více než 18 let.
- 2. Byl (a) jsem podrobně informován (a) o cílu studie, o jejích postupech, a o tom, co se ode mě očekává. Lékař pověřený prováděním studie mi vysvětlil očekávané přínosy a případná zdravotní rizika, která by se mohla vyskytnout během mé účasti ve studii a vysvětlil mi, jak bude postupovat při výskytu jejího nežádoucího průběhu. Beru na vědomí, že prováděná studie je výzkumnou činností. Pokud je studie randomizovaná, beru na vědomí pravděpodobnost náhodného zařazení do jednotlivých skupin lišících se léčbou.
- 3. Informoval (a) jsem lékaře pověřeného studií o všech lécích, které mé dítě užívalo v posledních 28 dnech, i o těch, které v současnosti užívá. Bude-li nějaký lék dítěti předepsán jiným lékařem, budu ho informovat o své účasti v klinické studii a bez souhlasu lékaře pověřeného touto studií ho nevezmu.
- 4. Budu při své terapii s terapeutem mého dítěte spolupracovat a v případě výskytu jakéhokoliv neobvyklého nebo nečekaného příznaku ho budu ihned informovat.
- 5. Po celou dobu studie a další 4 týdny po jejím ukončení nebude mé dítě dárcem krve.
- 6. Porozuměl (a) jsem tomu, že účast svého dítěte ve studii mohu kdykoliv přerušit či odstoupit, aniž by to jakkoliv ovlivnilo průběh mého dalšího léčení. Účast mého dítěte ve studii je dobrovolná.
- 7. Při zařazení do studie budou moje a mého dítěte osobní data uchována s plnou ochranou důvěrnosti dle platných zákonů ČR. Do původní zdravotní dokumentace dítěte budou moci na základě mého uděleného souhlasu nahlédnout za účelem ověření získaných údajů zástupci nezávislých etických komisí a zahraničních nebo místních kompetentních úřadů. Pro tyto případy je zaručena ochrana důvěrnosti mých osobních dat. Při vlastním provádění studie mohou být osobní údaje poskytnuty jiným než výše uvedeným subjektům pouze bez identifikačních údajů, to je anonymní data pod číselným kódem.Rovněž pro výzkumné a vědecké účely mohou být osobní údaje poskytnuty pouze bez identifikačních údajů (anonymní data) nebo s mým výslovným souhlasem.
- 8. S účastí mého dítěte ve studii není spojeno poskytnutí žádné odměny.
- 9. Porozuměl(a) jsem tomu, že jméno mého dítěte se nebude nikdy vyskytovat v referátech o této studii. Já pak naopak nebudu proti použití výsledků z této studie.

10. Převzal/a jsem podepsaný stejnopis tohoto informovaného souhlasu.

| Podpis pacienta: | Podpis lékaře pověřeného touto studií: |
|------------------|----------------------------------------|
| Datum: | Datum: |

### Reference

- 1. Chali F, Desseille C, Houdebine L, Benoit E, Rouquet T, Bariohay B, et al. Long-term exercise-specific neuroprotection in spinal muscular atrophy-like mice. J Physiol. 2016;594(7):1931-52.
- 2. Pera MC, Coratti G, Mazzone ES, Montes J, Scoto M, De Sanctis R, et al. Revised upper limb module for spinal muscular atrophy: 12 month changes. Muscle Nerve. 2019;59(4):426-30.
- 3. Carter GT, Abresch RT, Fowler WM, Jr., Johnson ER, Kilmer DD, McDonald CM. Profiles of neuromuscular diseases. Spinal muscular atrophy. Am J Phys Med Rehabil. 1995;74(5 Suppl):S150-9.
- 4. Lewelt A, Krosschell KJ, Stoddard GJ, Weng C, Xue M, Marcus RL, et al. Resistance strength training exercise in children with spinal muscular atrophy. Muscle Nerve. 2015;52(4):559-67.
- 5. Woo CJ, Maier VK, Davey R, Brennan J, Li G, Brothers J, 2nd, et al. Gene activation of SMN by selective disruption of lncRNA-mediated recruitment of PRC2 for the treatment of spinal muscular atrophy. Proc Natl Acad Sci U S A. 2017;114(8):E1509-e18.
- 6. Mazzone E, De Sanctis R, Fanelli L, Bianco F, Main M, van den Hauwe M, et al. Hammersmith Functional Motor Scale and Motor Function Measure-20 in non ambulant SMA patients. Neuromuscul Disord. 2014;24(4):347-52.
- 7. Jarman NF, Brooks T, James CR, Hooper T, Wilhelm M, Brismée JM, et al. Deep Neck Flexor Endurance in the Adolescent and Young Adult: Normative Data and Associated Attributes. Pm r. 2017;9(10):969-75.
- 8. Čapková K. Možnosti hipoterapie u dětských pacientů s dětskou mozkovou obrnu. . Čas Rehabilitace a fyzlékařství. 2016;2.
- 9. Cunha MC, Oliveira AS, Labronici RH, Gabbai AA. Spinal muscular atrophy type II (intermediary) and III (Kugelberg-Welander). Evolution of 50 patients with physiotherapy and hydrotherapy in a swimming pool. Arq Neuropsiquiatr. 1996;54(3):402-6.
- 1. Dunaway S, Montes J, McDermott MP, Martens W, Neisen A, Glanzman AM, et al. Physical therapy services received by individuals with spinal muscular atrophy (SMA). J Pediatr Rehabil Med. 2016;9(1):35-44.
- 2. Lewelt A, Krosschell KJ, Stoddard GJ, Weng C, Xue M, Marcus RL, et al. Resistance strength training exercise in children with spinal muscular atrophy. Muscle Nerve. 2015;52(4):559-67.
- 3. Montes J, Garber CE, Kramer SS, Montgomery MJ, Dunaway S, Kamil-Rosenberg S, et al. Single-Blind, Randomized, Controlled Clinical Trial of Exercise in Ambulatory Spinal Muscular Atrophy: Why are the Results Negative? J Neuromuscul Dis. 2015;2(4):463-70.
- 4. Mercuri E, Finkel RS, Muntoni F, Wirth B, Montes J, Main M, et al. Diagnosis and management of spinal muscular atrophy: Part 1: Recommendations for diagnosis, rehabilitation, orthopedic and nutritional care. Neuromuscul Disord. 2018;28(2):103-15.
- 5. Trenkle J, Brugman J, Peterson A, Roback K, Krosschell KJ. Filling the gaps in knowledge translation: Physical therapy recommendations for individuals with spinal muscular atrophy compared to standard of care guidelines. Neuromuscular Disorders. 2021;31(5):397-408.